CLINICAL TRIAL: NCT00703742
Title: A Neuroimaging and Epigenetic Investigation of Antidepressants in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kunming Medical University (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Yuqi Cheng, Vise director, psychiatry department, Kunming Medical University, Kunming Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Kunming MC
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Depression; Depression Secondary to Other Disease
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A,1 (Experimental): A: Escitalopram, 20 mg/day,8weeks
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — A,1: Escitalopram, oral, 20 mg/day, 8 weeks

SUMMARY:
The purpose of this study is:

1. to find out the structural or functional effects of selective serotonin reuptake inhibitors (SSRI) in major depressive disorder (MDD);
2. find special abnormalities in depression secondary to other disease, e.g., autoimmune disease like systemic lupus erythematosus (SLE).
3. find the relationship between the efficacy of antidepressant and the change of neuroimaging in MDD
4. to find possible predispose to MDD
5. to explore the DNA methylation status in depression;

DETAILED DESCRIPTION:
1. to explore the pathology of depression
2. to identify the difference between MDD and depression secondary to other disease ,especially autoimmune disease
3. to explore the effect of gene-environment interaction on the epigenetic regulation of the depression

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Major Depression or Dysthymia
* Age 18-65
* Physically healthy
* Drug-free

Exclusion Criteria:

* Body metal (e.g., wire stitches, screws in bones, stainless steel hips)
* History of Psychosis or Epilepsy
* Current (past six months) Substance Use Disorder (illicit drugs and/or alcohol)
* Bipolar I
* Need for wash-out from effective treatment in order to participate
* Pregnant
* High suicide risk
* Currently taking (within 2 weeks; 4 weeks for Fluoxetine) antidepressants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
change of fMRI after medication | baseline, 4 weeks, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xu Xiufeng, Study Director — Kunming Medical University
Locations (1):
- The First Affiliated Hospital of Kunming Medical College, Kunming, Yunnan, China

REFERENCES:
- [Derived] Chu Z, Yuan L, He M, Cheng Y, Lu Y, Xu X, Shen Z. Atrophy of bilateral nucleus accumbens in melancholic depression. Neuroreport. 2023 Jun 7;34(10):493-500. doi: 10.1097/WNR.0000000000001915. Epub 2023 May 31. PMID 37270840
- [Derived] Cheng Y, Xu J, Yu H, Nie B, Li N, Luo C, Li H, Liu F, Bai Y, Shan B, Xu L, Xu X. Delineation of early and later adult onset depression by diffusion tensor imaging. PLoS One. 2014 Nov 13;9(11):e112307. doi: 10.1371/journal.pone.0112307. eCollection 2014. PMID 25393297
- [Derived] Xu J, Cheng Y, Chai P, Lu Z, Li H, Luo C, Li X, Li L, Zhou Q, Chen B, Cao J, Xu X, Shan B, Xu L, Wen J. White-matter volume reduction and the protective effect of immunosuppressive therapy in systemic lupus erythematosus patients with normal appearance by conventional magnetic resonance imaging. J Rheumatol. 2010 May;37(5):974-86. doi: 10.3899/jrheum.090967. Epub 2010 Mar 15. PMID 20231206